CLINICAL TRIAL: NCT01403675
Title: Human Ovarian Autotransplantation Using Cryopreserved Ovarian Tissue in Women Treated for Cancer
Brief Title: Human Ovarian Autotransplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Kim, MD (Other)
Responsible Party: Sponsor-Investigator, Samuel Kim, MD, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11214
Record Dates: First submitted 2011-07-14; First posted 2011-07-27 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Ovarian Autotransplantation Using Cryopreserved Ovarian Tissue in Women Treated for Cancer
Keywords: women with cancer whose ovarian tissue has been collected and stored in liquid nitrogen before cancer therapy (surgery, chemotherapy, radiotherapy),; who are in remission (no recurrence of disease for 5 years),; who are in normal organ function and have no contraindication for surgery or pregnancy, and; who wish to restore ovarian function using stored ovarian tissue.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ovarian autotransplantation (Experimental)
  Interventions: Procedure: Ovarian autotransplantation

INTERVENTIONS:
Procedure: Ovarian autotransplantation — There are two ways to transplant the thawed ovarian tissue back into a woman's body. It can be put back inside the abdomen, close to the natural location of the ovaries, or the tissue can be put under the skin of the abdomen. After you have had the transplant, your hormone function will be tested every month. Each month, you will have a blood draw to measure hormones and an ultrasound to see how the tissue is growing. These monthly visits will continue until you have normal hormone levels. If the transplant is successful, it is expected that your hormones would return to normal in 3 - 7 months. If your hormone levels return and stay regular for three months, then Dr. Kim will talk to you about trying to get pregnant. The method of getting pregnant will depend on the type of transplantation surgery you had and your current medical condition. You will have weekly blood tests and other tests to determine the best way to get pregnant.

SUMMARY:
Chemotherapy can cause permanent damage to a woman's ovaries. Women who are cancer survivors may find that they are not able to produce female hormones, and they may not be able to have a child. Scientists are trying to find ways to help cancer survivors regain their hormonal function and possibly get pregnant, if they desire. Scientists have developed a method where ovarian tissue is removed and frozen before chemotherapy; then it is thawed and put back into the woman's body after she is cancer-free. Putting a woman's previously-frozen tissue back into her body is called ovarian autotransplantation.

Ovarian autotransplantation is a very new technique, and there have only been a small number of women who have had this procedure. So far, only five babies in the world have been born using this technique.

The purpose of this study is to learn more about ovarian autotransplantation. Scientists hope to find better ways to use this method to help a woman's ovaries start working again after chemotherapy. If the ovaries start working again, it might be possible to have a baby.

ELIGIBILITY:
Inclusion criteria:

* Adult women (age between 18 and 40) who stored the ovary before cancer therapy.
* Adult women who completed cancer therapy and are in remission.
* Adult women who desire to conceive and are ready to have a baby.

Exclusion criteria:

* Age under 18 or over 40 years old
* Women with a disease at high risk for ovarian metastasis (such as leukemia)
* Women with contraindication for surgery
* Women with contraindication for pregnancy
* Psychological instability to sustain pregnancy (diagnosed by a psychiatrist)
* Women who are HIV Positive

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2009-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Comparision of orthotopic and heterotopic autotransplantation | 2009-2015
  The main purpose of this study is to investigate restoration of ovarian function and fertility by autotransplantation of human ovarian tissue using heterotopic and orthotopic techniques

CONTACTS AND LOCATIONS:
Overall Officials: Sam Kim, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States